CLINICAL TRIAL: NCT04916522
Title: COHERENT - The COlchicine HypERtENsion Trial
Brief Title: The COlchicine HypERtENsion Trial
Acronym: COHERENT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Niklas Dyrby Johansen, Principal Investigator, MD, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COHERENT; 2020-004492-40 (EudraCT Number)
Record Dates: First submitted 2021-05-28; First posted 2021-06-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
Keywords: Inflammation; Vascular Stiffness; Pulse Wave Analysis; Blood Pressure; Echocardiography; Magnetic Resonance Imaging; Computed Tomography Angiography; Hypertrophy, Left Ventricular; Ventricular Function, Left; Endomyocardial Fibrosis; Atherosclerosis; Coronary Atherosclerosis; Colchicine; Cardiovascular Diseases; Heart Diseases; Randomized Controlled Trial
MeSH Terms: conditions — Hypertension; Inflammation; Hypertrophy, Left Ventricular; Endomyocardial Fibrosis; Atherosclerosis; Coronary Artery Disease; Cardiovascular Diseases; Heart Diseases | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental): Colchicine 0.5 mg once daily
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — 0.5 mg once daily
  Arms: Colchicine
Drug: Placebo — Once daily
  Arms: Placebo

SUMMARY:
The purpose of this study to investigate the effects of colchicine on measures of vascular and cardiac function in patients with hypertension.

DETAILED DESCRIPTION:
The study is an investigator-initiated, prospective, double-blind, placebo-controlled, randomized clinical trial investigating the effects of colchicine in patients with hypertension. The study population will consist of approximately 150 patients aged 18 years and above with a diagnosis of hypertension and in active treatment with at least 1 antihypertensive drug. Patients will be randomized to either low-dose colchicine treatment (0,5 mg once daily) or placebo. Treatment will continue for 6 months. Patients will be assessed by measurement of pulse wave velocity (PWV), office blood pressure, echocardiography, cardiac MRI, and blood samples at baseline and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Living address in the Capital Region of Denmark
2. Age >18 years
3. Diagnosed with hypertension
4. Treatment with 1 or more antihypertensive medications
5. Must fulfill at least one of the following high-risk criteria:

   1. Diagnosed with type 2 diabetes mellitus OR
   2. Treatment with lipid-lowering medication for dyslipidemia OR
   3. Treatment with 2 or more antihypertensive medications
6. Female patients should either not be of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing potential and practicing one of the following methods of contraception throughout the study and for 30 days after study completion: Hormonal contraception (oral contraceptives, contraceptive implant, injectable birth control, contraceptive patch, or vaginal ring) or intrauterine device
7. Patients will have given written, informed consent and are able and willing to comply with the requirements of the study protocol

Exclusion Criteria:

1. Colchicine treatment for another cause, e.g. gout
2. Allergy/hypersensitivity to colchicine
3. Known or suspected secondary hypertension, e.g. renal artery stenosis
4. Uncontrolled hypertension (systolic BP >180 mmHg or diastolic BP >110 mmHg)
5. Known other cardiovascular disease (judged by the investigator), e.g. ischemic heart disease, heart failure, significant valvular disease, arrhythmia, stroke, or peripheral artery disease
6. History of malignancy of any organ system excluding a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma, localized prostate cancer and/or localized carcinoma in situ of the cervix
7. Cirrhosis, chronic active hepatitis or other severe hepatic disease
8. Hemodialysis
9. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2
10. Systemic treatment with moderate or strong cytochrome P450 3A4 (CYP3A4) inhibitors or P-glycoprotein inhibitors
11. Anemia, thrombocytopenia or leucopenia defined as any of the following measurements within the last 3 months:

    1. Hemoglobin < 7 mmol/L
    2. Platelet count < 110 x 10^9/L
    3. White blood cell count < 3.0 x 10^9/L
12. Female patients who are pregnant, lactating, or considering becoming pregnant during the study or for 6 months after study completion
13. Significant drug or alcohol abuse during the last year
14. Current use of or plans to initiate chronic systemic steroid therapy during the study (topical or inhaled steroids are allowed)
15. Chronic inflammatory bowel disease (Crohn's disease or ulcerative colitis) or chronic diarrhea
16. Use of other investigational drugs within 30 days of the time of enrollment
17. Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in change in carotid-femoral pulse wave velocity at 6 months | 6 months

SECONDARY OUTCOMES:
Between-group difference in change in office-measured systolic blood pressure at 6 months | 6 months
Between-group difference in change in office-measured diastolic blood pressure at 6 months | 6 months
Between-group difference in change in left ventricular mass assessed by echocardiography at 6 months | 6 months
Between-group difference in change in left ventricular mass assessed by cardiac magnetic resonance imaging at 6 months | 6 months
Between-group difference in change in high sensitivity C-reactive protein at 6 months | 6 months
Between-group difference in change in high sensitivity Troponin I at 6 months | 6 months

OTHER OUTCOMES:
Between-group difference in change in office-measured pulse pressure at 6 months | 6 months
Between-group difference in change in central blood pressure assessed by pulse wave analysis at 6 months | 6 months
Between-group difference in change in augmentation index assessed by pulse wave analysis at 6 months | 6 months
Between-group difference in change in left ventricular septal wall thickness assessed by echocardiography at 6 months | 6 months
Between-group difference in change in left ventricular posterior wall thickness assessed by echocardiography at 6 months | 6 months
Between-group difference in change in left ventricular ejection fraction assessed by echocardiography at 6 months | 6 months
Between-group difference in change in E/A ratio assessed by echocardiography at 6 months | 6 months
Between-group difference in change in e' assessed by echocardiography at 6 months | 6 months
Between-group difference in change in E/e' assessed by echocardiography at 6 months | 6 months
Between-group difference in change in E/e'sr assessed by echocardiography at 6 months | 6 months
Between-group difference in change in left atrial volume assessed by echocardiography at 6 months | 6 months
Between-group difference in change in global longitudinal strain assessed by echocardiography at 6 months | 6 months
Between-group difference in change in myocardial work assessed by echocardiography at 6 months | 6 months
Between-group difference in change in aortic distensibility assessed by echocardiography at 6 months | 6 months
Between-group difference in change in aortic strain assessed by echocardiography at 6 months | 6 months
Between-group difference in change in left ventricular septal wall thickness assessed by cardiac magnetic resonance imaging at 6 months | 6 months
Between-group difference in change in left ventricular posterior wall thickness assessed by cardiac magnetic resonance imaging at 6 months | 6 months
Between-group difference in change in left ventricular ejection fraction assessed by cardiac magnetic resonance imaging at 6 months | 6 months
Between-group difference in change in left atrial volume assessed by cardiac magnetic resonance imaging at 6 months | 6 months
Between-group difference in change in myocardial fibrosis assessed by cardiac magnetic resonance imaging at 6 months | 6 months
Between-group difference in change in myocardial inflammation assessed by cardiac magnetic resonance imaging at 6 months | 6 months
Between-group difference in change in tumor necrosis factor alpha at 6 months | 6 months
Between-group difference in change in pro B-type natriuretic peptide at 6 months | 6 months
Between-group difference in change in interleukin-1 beta at 6 months | 6 months
Between-group difference in change in interleukin-6 at 6 months | 6 months
Between-group difference in change in interleukin-10 at 6 months | 6 months
Between-group difference in change in interleukin-17 at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Dyrby Johansen, MD, Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Cardiovascular Non-Invasive Imaging Research Laboratory, Department of Cardiology, Herlev and Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes